CLINICAL TRIAL: NCT04416100
Title: Development of Interstitial Lung Disease (ILD) in Patients With Severe SARS-CoV-2 Infection
Brief Title: Development of Interstitial Lung Disease (ILD) in Patients With Severe SARS-CoV-2 Infection (COVID-19)
Acronym: CovILD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 20200429-2255
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-05

CONDITIONS: Covid-19; Pulmonary Fibrosis
MeSH Terms: conditions — COVID-19; Pulmonary Fibrosis | interventions — Respiratory Function Tests; Diagnostic Imaging; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of peripheral blood will be done in the context of a routine blood draw in all study participants (in addition for immunofibrotic phenotyping) at our study centre at indicated time-points.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Pulmonary function tests — Spirometry or plethysmography, measurement of diffusion capacity
Diagnostic Test: Imaging — HRCT and echocardiography as scheduled within routine clinical examinations
Biological: Blood sampling — Standard laboratory test as part of routine clinical examination and collection of peripheral blood for immunofibrotic phenotyping

SUMMARY:
COVID-19, the infectious disease caused by the novel coronavirus SARS-CoV-2, currently poses a global economic, social, political and medical challenge. The virus originated in December 2019 in Wuhan, China, and has spread rapidly around the world. Currently, European countries, including Austria, are severely affected.The most common computed tomographic changes in acute lung injury include bilateral and subpleural milk glass opacity, consolidation in lower lobes, or both. In the intermediate phase of the infection (4-14 days after the onset of symptoms) a so-called "crazy paving" may occur. The most prominent radiological changes occur around day 10, followed by gradual resolution, which begins two weeks after the onset of symptoms.

Given the phylogenetic relationship between SARS-CoV-1 and SARS-CoV-2, the similar clinical course in severe cases and overlapping CT patterns in the acute setting, persistent radiological and pulmonary functional changes in survivors are conceivable. It is also conceivable that a proportion of survivors will develop progressive ILD, either due to viral or ventilator-induced alveolar damage, or both.

Here, the investigators intend to investigate COVID-19 survivors through clinical examinations, functional lung examinations, HR-CT scans, and by determining the "immunofibrotic" pattern in peripheral mononuclear cells (PBMCs) 1, 3, and 6 months after discharge.

DETAILED DESCRIPTION:
COVID-19, the infectious disease caused by the novel coronavirus SARS-CoV-2, currently poses a global economic, social, political and medical challenge. The virus originated in December 2019 in Wuhan, China, and has spread rapidly around the world. Currently, European countries, including Austria, are severely affected. In January 2020, the World Health Organisation declared a "Public Health Event of International Concern" and since 11 March 2020 COVID-19 has been classified as a pandemic. Overall mortality rates vary widely, ranging from 0.5 to 7%. These highly depend on the stringency of the tests in a particular region and the age of the patients with higher mortality rates in older people. The majority of patients show only mild symptoms with fever and/or cough, and it is even believed that there is a significant proportion of untested asymptomatic carriers that can transmit the virus to other people. 26 to 33% of in-patients have been admitted to intensive care due to a severe lung disease. Of these, 2.5 to 10% required invasive mechanical ventilation and 15 to 22% of these patients died in hospital, indicating the potential risk to public health. As a result, the current global death toll from COVID-19 already exceeds 37,000 people on 31 March 2020.

In the SARS-CoV-1 outbreak of 2003, clinical course was characterized by fever, myalgia and other systemic symptoms, which generally improved after a few days, followed by a second phase with recurrence of fever, oxygen saturation and imaging progression of pneumonia, similar to that experienced by severely affected patients in the current pandemic. Importantly, a significant number of patients infected with SARS-CoV-1 suffered acute respiratory failure (ARDS) requiring invasive ventilatory support. The pulmonary pathology of fatal SARS cases was dominated by diffuse alveolar damage (DAD), epithelial cell proliferation, an increase in macrophages in the lung and extensive consolidation, but features of bronchiolitis obliterans and organizing pneumonia were also noted. In addition, survivors of severe SARS-CoV-1 infection showed significant functional and radiological changes in the lungs even 6 months after infection.

In the current SARS-CoV-2 pandemic, the most common computed tomographic changes in acute lung injury include bilateral and subpleural milk glass opacity, consolidation in lower lobes, or both. In the intermediate phase of the infection (4-14 days after the onset of symptoms) a so-called "crazy paving" may occur. The most prominent radiological changes occur around day 10, followed by gradual resolution, which begins two weeks after the onset of symptoms.

Given the phylogenetic relationship between SARS-CoV-1 and SARS-CoV-2, the similar clinical course in severe cases and overlapping CT patterns in the acute setting, persistent radiological and pulmonary functional changes in survivors are conceivable. It is also conceivable that a proportion of survivors will develop progressive ILD, either due to viral or ventilator-induced alveolar damage, or both.

Here, the investigators intend to investigate COVID-19 survivors through clinical examinations, functional lung examinations, HR-CT scans, and by determining the "immunofibrotic" pattern in peripheral mononuclear cells (PBMCs) 1, 3, and 6 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients ≥ 18 years.
* Confirmed infection with SARS-CoV-2 according to the definition of the Austrian Federal Ministry of Social Affairs, Health, Care and Consumer Protection
* Signed and dated declaration of consent by the patient according to ICH-GCP Guidelines.

Exclusion Criteria:

* Female and male patients < 18 years
* Pregnancy
* Dementia
* Declaration of consent by the patient according to ICH-GCP Guidelines not signed
* Incapacitated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients discharged from hospital or outpatients referred to our Outpatient Department of Pneumology at the University Hospital of Innsbruck because of persistent respiratory symptoms in recovery phase will be followed up. Diagnosis of COVID-19 must have been ensured by nasopharyngeal and oropharyngeal swabs.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-04-29 (Actual); Primary Completion 2022-04-28 (Estimated); Study Completion 2022-04-28 (Estimated)

PRIMARY OUTCOMES:
Pattern of pulmonary abnormalities in SARS-CoV2 infected patients after 1 month | 1 month
  Define the frequency of ILD and pulmonary vascular disease in SARS-CoV-2 infected patients with a severe/prolonged Course (inhospital stay, either on the normal ward or ICU), with and without oxygen supplementation, non-invasive or invasive ventilation) at 1 month after discharge or diagnosis of COVID-19 disease by the use of HR-CT.
Pattern of pulmonary abnormalities in SARS-CoV2 infected patients after 3 months | 3 months
  Define the frequency of ILD and pulmonary vascular disease in SARS-CoV-2 infected patients with a severe/prolonged Course (inhospital stay, either on the normal ward or ICU), with and without oxygen supplementation, non-invasive or invasive ventilation) at 3 months after discharge or diagnosis of COVID-19 disease by the use of HR-CT
Pattern of pulmonary abnormalities in SARS-CoV2 infected patients after 6 months | 6 months
  Define the frequency of ILD and pulmonary vascular disease in SARS-CoV-2 infected patients with a severe/prolonged Course (inhospital stay, either on the normal ward or ICU), with and without oxygen supplementation, non-invasive or invasive ventilation) at 6 months after discharge or diagnosis of COVID-19 disease by the use of HR-CT

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Tancevski, Doz. Dr., Principal Investigator — Medical University Innsbruck, Department Internal Medicine II
Locations (1):
- Medical University of Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rass V, Tymoszuk P, Sahanic S, Heim B, Ausserhofer D, Lindner A, Kofler M, Mahlknecht P, Boehm A, Hufner K, Pizzini A, Sonnweber T, Kurz K, Pfeifer B, Kiechl S, Peball M, Kindl P, Putnina L, Fava E, Djamshidian A, Huber A, Wiedermann CJ, Sperner-Unterweger B, Woll E, Beer R, Schiefecker AJ, Bellmann-Weiler R, Bachler H, Tancevski I, Pfausler B, Piccoliori G, Seppi K, Weiss G, Loffler-Ragg J, Helbok R. Distinct smell and taste disorder phenotype of post-acute COVID-19 sequelae. Eur Arch Otorhinolaryngol. 2023 Nov;280(11):5115-5128. doi: 10.1007/s00405-023-08163-x. Epub 2023 Sep 5. PMID 37670171
- [Derived] Hufner K, Tymoszuk P, Sahanic S, Luger A, Boehm A, Pizzini A, Schwabl C, Koppelstatter S, Kurz K, Asshoff M, Mosheimer-Feistritzer B, Pfeifer B, Rass V, Schroll A, Iglseder S, Egger A, Woll E, Weiss G, Helbok R, Widmann G, Sonnweber T, Tancevski I, Sperner-Unterweger B, Loffler-Ragg J. Persistent somatic symptoms are key to individual illness perception at one year after COVID-19 in a cross-sectional analysis of a prospective cohort study. J Psychosom Res. 2023 Jun;169:111234. doi: 10.1016/j.jpsychores.2023.111234. Epub 2023 Mar 17. PMID 36965396
- [Derived] Nagele F, Graber M, Hirsch J, Polzl L, Sahanic S, Fiegl M, Hau D, Engler C, Lechner S, Stalder AK, Mertz KD, Haslbauer JD, Tzankov A, Grimm M, Tancevski I, Holfeld J, Gollmann-Tepekoylu C. Correlation between structural heart disease and cardiac SARS-CoV-2 manifestations. Commun Med (Lond). 2022 Nov 11;2(1):142. doi: 10.1038/s43856-022-00204-6. PMID 36369278
- [Derived] Sviridenko A, Boehm A, di Santo G, Uprimny C, Nilica B, Fritz J, Giesel FL, Haberkorn U, Sahanic S, Decristoforo C, Tancevski I, Widmann G, Loeffler-Ragg J, Virgolini I. Enhancing Clinical Diagnosis for Patients With Persistent Pulmonary Abnormalities After COVID-19 Infection: The Potential Benefit of 68 Ga-FAPI PET/CT. Clin Nucl Med. 2022 Dec 1;47(12):1026-1029. doi: 10.1097/RLU.0000000000004437. Epub 2022 Oct 15. PMID 36257062
- [Derived] Sonnweber T, Tymoszuk P, Sahanic S, Boehm A, Pizzini A, Luger A, Schwabl C, Nairz M, Grubwieser P, Kurz K, Koppelstatter S, Aichner M, Puchner B, Egger A, Hoermann G, Woll E, Weiss G, Widmann G, Tancevski I, Loffler-Ragg J. Investigating phenotypes of pulmonary COVID-19 recovery: A longitudinal observational prospective multicenter trial. Elife. 2022 Feb 8;11:e72500. doi: 10.7554/eLife.72500. PMID 35131031
- [Derived] Sonnweber T, Sahanic S, Pizzini A, Luger A, Schwabl C, Sonnweber B, Kurz K, Koppelstatter S, Haschka D, Petzer V, Boehm A, Aichner M, Tymoszuk P, Lener D, Theurl M, Lorsbach-Kohler A, Tancevski A, Schapfl A, Schaber M, Hilbe R, Nairz M, Puchner B, Huttenberger D, Tschurtschenthaler C, Asshoff M, Peer A, Hartig F, Bellmann R, Joannidis M, Gollmann-Tepekoylu C, Holfeld J, Feuchtner G, Egger A, Hoermann G, Schroll A, Fritsche G, Wildner S, Bellmann-Weiler R, Kirchmair R, Helbok R, Prosch H, Rieder D, Trajanoski Z, Kronenberg F, Woll E, Weiss G, Widmann G, Loffler-Ragg J, Tancevski I. Cardiopulmonary recovery after COVID-19: an observational prospective multicentre trial. Eur Respir J. 2021 Apr 29;57(4):2003481. doi: 10.1183/13993003.03481-2020. Print 2021 Apr. PMID 33303539
- [Derived] Sonnweber T, Boehm A, Sahanic S, Pizzini A, Aichner M, Sonnweber B, Kurz K, Koppelstatter S, Haschka D, Petzer V, Hilbe R, Theurl M, Lehner D, Nairz M, Puchner B, Luger A, Schwabl C, Bellmann-Weiler R, Woll E, Widmann G, Tancevski I, Judith-Loffler-Ragg, Weiss G. Persisting alterations of iron homeostasis in COVID-19 are associated with non-resolving lung pathologies and poor patients' performance: a prospective observational cohort study. Respir Res. 2020 Oct 21;21(1):276. doi: 10.1186/s12931-020-01546-2. PMID 33087116